CLINICAL TRIAL: NCT06904417
Title: Effect of the Feldenkrais Method on Enhancing Postural Control in Patients with Diabetic Polyneuropathy
Brief Title: Effect of Feldenkrais Method in Enhancing Postural Control for Patients with Diabetic Polyneuropathy
Acronym: FeM
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Islam Hassan Fayed, Physiotherapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005646
Record Dates: First submitted 2025-02-05; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2024-12

CONDITIONS: Diabetic Polyneuropathy
Keywords: Feldenkrais Method; Postural Control; Diabetic Polyneuropathy
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Intervention Model Description: The Feldenkrais-based intervention consisted of guided awareness exercises aimed at improving movement patterns, proprioception, and postural control. Sessions were conducted twice weekly for 12 weeks, with each session lasting approximately 45 minutes.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The Feldenkrais-based intervention (Experimental): this group recieve The Feldenkrais-based intervention consisted of guided awareness exercises
  Interventions: Other: The Feldenkrais-based intervention
- a conventional balance training program (Active Comparator): The control group participated in a conventional balance training program consisting of static and dynamic balance exercises, gait training, and strength-building activities, matched for session frequency and duration

INTERVENTIONS:
Other: The Feldenkrais-based intervention — The Feldenkrais-based intervention consisted of guided awareness exercises aimed at improving movement patterns, proprioception, and postural control. Sessions were conducted twice weekly for 12 weeks, with each session lasting approximately 45 minutes
  Arms: The Feldenkrais-based intervention
Other: conventional balance training program — a conventional balance training program consisting of static and dynamic balance exercises, gait training, and strength-building activities, matched for session frequency and duration

SUMMARY:
Background: Postural Control is a major complication of polyneuropathy, affecting patients suffering from diabetes mellitus. Purpose: To examine the effect of the Feldenkrais Method on dynamic balance, limits of stability and fear of falling in adults aged 45 to 60 years with diabetic polyneuropathy in the short and mid-term. Methods: A single-blinded, parallel, multicentric randomized control trial was conducted in two health centers. Adults aged 45 to 60 years with diabetic polyneuropathy and a history of falls or dynamic balance dysfunction were recruited from hospital databases and randomly assigned to either the study or control group. The study group received 16 sessions of Feldenkrais-based sensorimotor training. Both groups received diabetic foot care instructions and traditional balance exercises. Outcomes were measured at 3 and 6-month follow-up intervals. Dynamic balance was assessed using the Timed Up and Go (TUG) Test, limits of stability using Biodex and fear of falling with the Falls Efficacy Scale (FES).

ELIGIBILITY:
Inclusion Criteria:

* Individuals must have a diagnosis of Diabetic Polyneuropathy (DPN), confirmed by clinical examination and electrophysiological testing.
* Participants must have stable glycemic control for at least three months prior to enrollment.
* Individuals must be able to walk independently, with or without the use of an assistive device.

Exclusion Criteria:

* Individuals with severe visual or vestibular impairments are excluded from participation.
* Participants with significant musculoskeletal disorders affecting gait are not eligible.
* Individuals with severe cardiovascular or respiratory conditions are excluded.
* Participants with cognitive impairments that prevent active participation are not eligible.
* Individuals currently engaged in structured physical therapy or balance training programs are excluded.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-03-30 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Dynamic Balance | From enrollment to the end of treatment at 12 weeks
  Assessed using the Timed Up and Go Test, which measures the time taken to stand from a seated position, walk three meters, turn around, walk back, and sit down.
Postural Control | From enrollment to the end of treatment at 12 weeks
  Evaluated using the Biodex Balance System, which measures limits of stability and sway index
Fear of Falling | From enrollment to the end of treatment at 12 weeks
  Assessed using the Falls Efficacy Scale, a self-reported measure of confidence in performing daily activities without falling.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No